CLINICAL TRIAL: NCT00459784
Title: How to Reach Evidence Based Practice in Diagnostic Assessment and Management of Dementia by General Practitioners and Primary Care Nurses? The Effectiveness of an EASYcare Based Educational Program.
Brief Title: Implementation Study of Dementia Guidelines in Primary Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: County of Gelderland (Unknown); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Health Valley, Netherlands (Network); Stichting Thuiszorgorganisatie Midden-Gelderland (Unknown); Stichting Thuiszorgorganisatie Mawe Rivierenland (Unknown); Sensire Winterwijk (Unknown); Kruiswerk West Veluwe (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: EASYcareGIDS study
Record Dates: First submitted 2007-04-12; First posted 2007-04-13 (Estimated); Last update posted 2007-04-13 (Estimated); Status verified 2007-04

CONDITIONS: Dementia
Keywords: Improvement; Dementia early diagnosis; Dementia management; Primary care
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Dementia Training Program

SUMMARY:
The purpose of this study is to determine whether a specially developed Dementia Training Program for duos of general practitioners and primary care nurses is able to increase the number dementia diagnoses in elderly people living in the community and increase the adherence to clinical dementia guidelines

DETAILED DESCRIPTION:
Background Early diagnosis of dementia benefits both patient and caregiver. Nevertheless, dementia in primary care is currently under-diagnosed in developed countries. In several countries educational interventions were developed to improve dementia diagnosis and management in primary care. Some of these interventions were successful in increasing the number of dementia diagnoses and in changing attitudes and knowledge of health care staff. However, none of these interventions focussed on collaboration between GPs and nurses in dementia care. We developed a Dementia Training Program (DTP) aimed at stimulating collaboration in dementia primary care. We expect it to increase the number of cognitive assessments and dementia diagnoses, as well as to improve attitudes and knowledge of GPs and nurses.

Methods/Design The DTP is a complex educational intervention and consists of 2 workshops, a coaching program, and case-based consultations either face-to-face or by phone or e-mail, access to an internet forum, and a Computerized Clinical Decision Support System on dementia diagnostics and management. 100 duos of GPs and nurses will be recruited, from which 2/3 will be allocated to the intervention group and 1/3 to the control group. The effects of implementation of the DTP will be studied in an assessor blinded cluster-randomised controlled trial. Primary outcomes are the number of cognitive assessments and dementia diagnosis in a period of 9 months, starting after workshop participation of the duos. Secondary outcomes are measured on GP and nurse level: rate of adherence to national guidelines for dementia diagnosis, attitude, confidence and knowledge regarding dementia diagnosis and management; on patient level: number of emergency calls, visits and consultations and patient satisfaction; and on caregiver level: informal caregiver burden and satisfaction. Data will be collected from GPs' electronic medical dossiers, self registration forms and questionnaires. Statistical analysis will be performed by using MANOVA-method. Also, exploratory analyses will be performed, in order to gain insight into barriers and facilitators for implementation and the causal relations between the rate of success of the intervention components and the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* GP and practice or district nurse must participate as a duo

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2006-11; Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
Number of dementia diagnoses and cognitive assessments during 9 months

SECONDARY OUTCOMES:
Accuracy tot dementia guidelines, GP and nurse knowlegde and attitude and competence regarding dementia. Patient satisfaction, caregiver burden and satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Olde Rikkert, Prof, MD, Study Director — Alheimer Centre Nijmegen, the Netherlands
Locations (1):
- Geriatrie 925, Postbus 9101, Nijmegen, Netherlands

REFERENCES:
- [Derived] Perry M, Draskovic I, van Achterberg T, Borm GF, van Eijken MI, Lucassen P, Vernooij-Dassen MJ, Olde Rikkert MG. Can an EASYcare based dementia training programme improve diagnostic assessment and management of dementia by general practitioners and primary care nurses? The design of a randomised controlled trial. BMC Health Serv Res. 2008 Apr 2;8:71. doi: 10.1186/1472-6963-8-71. PMID 18384675